CLINICAL TRIAL: NCT02482623
Title: The Dementia Symptom Management at Home Program: A Bundled Interprofessional Intervention to Improve Dementia Patient-Caregiver Dyad Quality of Care and Quality of Life Through Home Healthcare.
Brief Title: The Dementia Symptom Management at Home Program
Acronym: DSM-H
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of study site
Sponsor: New York University (Other)
Collaborators: Visiting Nurse Service of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: i14-01960
Record Dates: First submitted 2015-06-23; First posted 2015-06-26 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2018-09

CONDITIONS: Dementia
Keywords: Dementia; neuropsychiatric symptoms; implementation science; depression; pain
MeSH Terms: conditions — Dementia; Depression; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dyads in this arm will receive care provided by an interprofessional team trained through the DSM-H to provide patient/caregiver-centered dementia care through home healthcare.
  Interventions: Behavioral: Dementia Symptom Management at Home Program
- Control (No Intervention): Dyads in this arm will receive usual care provided in the home healthcare setting.

INTERVENTIONS:
Behavioral: Dementia Symptom Management at Home Program — The DSM-H is a multi-modal interprofessional intervention that includes: 1. intensive training of clinician mentors; 2. disseminated online training for Registered Nurses, Physical Therapists, Occupational Therapists; 3. implementation of evidence-based care plans, assessment instruments, and teaching handouts.
  Other Names: DSM-H
  Arms: Intervention

SUMMARY:
Persons with dementia and their caregivers are often cared for in the community through home healthcare (HHC). While these patients and their caregivers need significant help and often have difficulty maintaining their quality of life, home healthcare clinicians are often unprepared to care for this population. This study will therefore examine the ability of an integrated, multi-pronged evidence-based practice intervention for home healthcare registered nurses, occupational therapists and physical therapists, the DSM-H, to improve the quality of care and quality of life for persons with dementia and their family caregiver. The investigators will enroll persons with dementia and their family caregiver upon admission to the HHC agency and examine their quality of life over 60 days following admission, comparing those who receive the intervention to those who serve as controls.

DETAILED DESCRIPTION:
The Dementia Symptom Management at Home (DSM-H) Program is an integrated bundled implementation science intervention to improve interprofessional care in home healthcare (HHC). It consists of training, assessment instruments, patient-caregiver centered care plans and workflow changes. The investigators will perform a cluster randomized controlled clinical trial at a single, urban, non-profit HHC agency, randomizing care teams to either be trained in performing the intervention or serve as controls. The aims of this program are to examine the efficacy of this program to:

Aim 1: Measure the effects of DSM-H on pain, neuropsychiatric symptoms, and caregiver rated QOL in the person with dementia receiving HHC.

Aim 2: Assess the effects of DSM-H on QOL, burden and depression for the informal caregiver of persons with dementia receiving HHC.

Aim 3: Assess the effects of DSM-H on the number of emergency room visits and hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* patient-caregiver dyad admitted to the HHC agency
* Patients must be 65 or older and speak English and/or Spanish.
* Patient must have an informal caregiver who is at least 18 years old and spends at least 8 hours per week with the patient.
* Patients must score greater than 4 on the cognitive subscale of the Healthy Aging Brain Care Monitor signifying at least mild impairment

Exclusion Criteria:

* Patients with concomitant axis I disorders other than dementia, depression, adjustment disorders, sleep disorders.
* Patients being seen only in the behavioral health unit without another skilled need.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Person With Dementia Quality of Life | 60 Days
  Quality of Life in Alzheimer's Disease survey instrument
Caregiver Quality of Life | 60 Days
  Caregiver Targeted Quality of Life survey instrument

SECONDARY OUTCOMES:
Person with Dementia Pain | 60 days
  Pain Assessment in Advanced Dementia or Brief Pain Inventory survey instrument
Person with Dementia Neuropsychiatric Symptom Burden | 60 days
  Healthy Aging Brain Care Monitor survey instrument
Caregiver Depression | 60 days
  Public Health Questionnaire-9 survey instrument
Person with Dementia ER Visits | 30, 60 days
  Resource Utilization Inventory survey instrument
Person with Dementia Hospital Admissions | 30, 60 days
  Resource Utilization Inventory survey instrument
Person with Dementia Functional Status | 60 days
  Katz Activities of Daily Living and Lawton Instrumental Activities of Daily Living assessments

CONTACTS AND LOCATIONS:
Overall Officials: Abraham A Brody, RN, PhD, GNP-BC, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - The New Jewish Home, New York, New York
  - New York University College of Nursing, New York, New York